CLINICAL TRIAL: NCT01982266
Title: A Prospective, Multicenter, Single Arm Feasibility Study of the Safety and Performance of GRADION™ Hip Total Cartilage Replacement (TCR)™ in the Treatment of Degenerative Joint Disease of the Hip
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device failure
Sponsor: Biomimedica, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP052
Record Dates: First submitted 2013-11-01; First posted 2013-11-13 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Degenerative Joint Disease of the Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GRADION™ Hip Total Cartilage Replacement (TCR)™ (Experimental)
  Interventions: Device: GRADION™ Hip Total Cartilage Replacement (TCR)™

INTERVENTIONS:
Device: GRADION™ Hip Total Cartilage Replacement (TCR)™

SUMMARY:
This is a prospective, multicenter, single arm feasibility study of the safety and performance of the GRADION™ Hip Total Cartilage Replacement (TCR)™ in patients who require cartilage replacement.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip surgery for Noninflammatory Degenerative Joint Disease (NIDJD) such as osteo/degenerative arthritis, and is indicated for cartilage replacement
* Skeletally mature or at least 18 years of age and has normal anatomy
* Patient signs the Informed Consent form
* Failed medical management
* There will be size limitations on patients also - available size range is 46mm-54mm.

Exclusion Criteria:

* Allergic to polyether urethane, sodium polyacrylate, bone cement or any of its components
* Previous fusion, acute femoral neck fracture and/or above knee amputation
* Revision of any previous hip procedure
* Slipped capital femoral epiphysis (SCFE)
* Rheumatoid arthritis
* AVN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Adverse events | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Arnhem, Arnhem, Netherlands